CLINICAL TRIAL: NCT06180083
Title: Single Dose Bioequivalence Study of Azelastine Hydrochloride/Fluticasone Propionate 137microgram/50 Microgram Nasal Spray and DYMISTA Nasal Spray in Healthy Adult Human Subjects
Brief Title: Bioequivalence Study of Azelastine Hydrochloride/ Fluticasone Propionate 137 Microgram/50 Microgram Nasal Spray and Dymista Nasal Spray
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B01728
Record Dates: First submitted 2023-12-09; First posted 2023-12-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Seasonal Allergic Rhinitis; Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial | interventions — azelastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azelastine Hydrochloride/ Fluticasone propionate nasal spray (Experimental): Azelastine Hydrochloride/ Fluticasone propionate 137 microgram/50 microgram nasal spray
  Interventions: Drug: Azelastine Hydrochloride/ Fluticasone propionate nasal spray; Drug: 'DYMISTA' NASAL SPRAY
- 'DYMISTA' Nasal Spray (Active Comparator): 'DYMISTA' (Azelastine Hydrochloride/ Fluticasone Propionate) Nasal Spray 137 microgram/50 microgram
  Interventions: Drug: Azelastine Hydrochloride/ Fluticasone propionate nasal spray; Drug: 'DYMISTA' NASAL SPRAY

INTERVENTIONS:
Drug: Azelastine Hydrochloride/ Fluticasone propionate nasal spray — A single dose [four sprays (two sprays in each nostril)] of Azelastine HCL/ Fluticasone Propionate 137 mcg/50 mcg Nasal Spray
Drug: 'DYMISTA' NASAL SPRAY — A single dose [four sprays (two sprays in each nostril)] of 'DYMISTA' (AZELASTINE HYDROCHLORIDE/ FLUTICASONE PROPIONATE) NASAL SPRAY 137 Microgram/50 Microgram

SUMMARY:
Single dose (four sprays) bioequivalence study of Azelastine Hydrochloride/ Fluticasone Propionate 137 microgram/50 microgram Nasal Spray and 'DYMISTA' (Azelastine Hydrochloride/Fluticasone Propionate) Nasal Spray 137 microgram/50 microgram in healthy adult human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45 years old, both inclusive.
* Gender: Male and/or non-pregnant, non-lactating female.

  1. Female of childbearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days prior to first dosing day. They used an acceptable form of contraception.
  2. For female of childbearing potential, acceptable forms of contraception included the following:

  i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remained in place during the study period, or ii. Barrier methods containing or used in conjunction with a spermicidal agent, or iii. Surgical sterilization or iv. Practiced sexual abstinence throughout the course of the study c)Female were not considered of childbearing potential in case one of the following was reported and documented on the medical history: i. Postmenopausal with spontaneous amenorrhea for at least one year, or ii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iii. Total hysterectomy and an absence of bleeding for at least 3 months.
* BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value were rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
* No nasal abnormalities.
* Non-smokers and non-tobacco users (i.e. had no past history of smoking and tobacco consuming for at least one year prior to study).
* The subject was willing to undergo the necessary pre- & post- medical examinations set by this study.
* Was able to communicate effectively with study personnel.
* Was able to understand and willing to provide written informed consent to participate in the study.
* All volunteers were judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which included:

  1. A physical examination (clinical examination) with no clinically significant finding.
  2. Results within normal limits or clinically non-significant for the following tests:

Hematology, Biochemistry, Urinalysis, Immunological Tests, Serum (β-HCG) pregnancy test (for female of child bearing potential)

Exclusion Criteria:

* History of allergic responses to Azelastine and Fluticasone Propionate or other related drugs, or any of its formulation ingredients.
* Had significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG, nasal examination [examination include (1) external nose but not limited to size and shape, obvious swellings or deformity, scars or skin changes and redness or discharge and (2) nasal cavity for but not limited to nasal septum, turbinates, entire nasal cavity for rhinitis, oedematous and inflamed mucosa, polyps or any other abnormalities and presence of any foreign bodies], Peak Nasal Inspiratory Flow measurement, chest X-ray recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* Any disease or condition like diabetes, psychosis or others, which compromised the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, Central nervous system or any other body system.
* History or presence of bronchial asthma.
* Used any hormone replacement therapy within 3 months prior to the first dose of study medication.
* A depot injection or implant of any drug within 3 months prior to the first dose of study medication.
* Used CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://drug-interactions.medicine.iu.edu/MainTable.aspx).
* History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* A positive hepatitis screen (includes subtypes B & C).
* A positive test result for HIV antibody and / or syphilis (RPR).
* Volunteers who had received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication or who had participated in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the first dose of study medication, whichever was greater.
* Volunteers who had donated blood within 80 days (excluding volume drawn at screening for this study) prior to first dose of study medication.
* Intolerance to venipuncture
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, contraindicated the volunteer's participation in this study.
* Institutionalized volunteers.
* Used any prescribed medications (including ritonavir, cobicistat & CNS depressants) within 14 days prior to the first dose of study medication.
* Used any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
* Used grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
* Ingested of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeinecontaining sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
* Ingested any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
* Volunteer had any illness since screening visit.
* Volunteer had any relevant disease including seasonal and perennial allergic rhinitis, asthma during screening.
* Volunteer had clinically relevant structural nasal abnormalities including deviated nasal septum, and upper respiratory tract infection within two weeks prior to the start of the study.
* Volunteer took steroids or any antihistamines or any drug related to allergic medication within 1 month prior to the dose of study medication.
* Volunteer who was not ready to remove Nasal jewelry prior to enrollment in the study
* Presence of nose piercings, which affected spray inhalation dosing and increase the deposition of the study drug in the nose.
* Presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis, or other eye infection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration(Cmax) | 120 hours
  The 90% confidence interval of the relative mean (geometric least square mean) of the test to reference product for Ln-transformed Pharmacokinetic parameters Cmax was to be within 80.00% to 125.00%
Area under the plasma concentration versus time curve from the zero time point to the last quantifiable concentration (AUCt) | 120 hours
  The 90% confidence intervals of the relative mean (Geometric least square mean) of the test to reference formulation for Ln-transformed AUCt was to be within 80.00% to 125.00%.
  bioequivalence.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time zero to infinity (AUCi) | 120 hours
  Descriptive statistics
Time of the maximum measured plasma concentration (Tmax) | 120 hours
  Descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No